CLINICAL TRIAL: NCT00150007
Title: Measurement of Patient Reported Outcomes in Renal Transplant Patients With and Without Gastrointestinal (GI) Symptoms (PROGIS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A2407
Record Dates: First submitted 2005-08-26; First posted 2005-09-08 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2011-11

CONDITIONS: Kidney Maintenance Transplant
Keywords: Kidney, maintenance transplant, GI complaints, patient reported outcome

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

SUMMARY:
The purpose of this study is to assess the impact that GI complaints have on patient reported outcomes in renal transplant recipients and to determine if there is improvement in patient reported outcomes when patients are converted to a EC-MPS-based immunosuppressive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Received kidney transplant at least 1 month prior to study enrollment;
* Receiving immunosuppressive regimen that includes MMF for at least 2 weeks prior to study enrollment;
* Eligible to convert to EC-MPS because of GI complaints OR not currently experiencing GI complaints and stable on current immunosuppressive regimen;
* At least 18 years of age;
* Willing to provide written informed consent; and
* Able to meet all study requirements including completing paper questionnaires and completing two study visits.

Exclusion Criteria:

* GI symptoms assumed or known not to be caused by MPA therapy (e.g. oral biphosphonates induced, infectious diarrhea);
* Acute rejection < 1 week prior to study enrollment;
* Woman of child-bearing potential who is planning to become pregnant or is pregnant and/or lactating who is unwilling to use effective means of contraception;
* Presence of psychiatric illness (i.e., schizophrenia, major depression) that, in the opinion of the site investigator, would interfere with study requirements;
* Undergoing acute medical intervention or hospitalization;
* Any other medical condition that, in the opinion of the site investigator based on recall or chart review, would interfere with completing the study, including but not limited to, visual problems or cognitive impairment
* Receiving any investigational drug or have received any investigational drug within 30 days prior to study enrollment.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 335
Dates: Start 2004-06; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Improvement in Gastro intestinal (GI) symptom severity and health-related quality of life (HRQoL) in patients with GI complaints who are converted from mycophenolate mofetil (MMF) to enteric-coated mycophenolate sodium (EC-MPS)

SECONDARY OUTCOMES:
Impact of GI symptoms on patients' perceptions of symptom severity, GI-specific HRQoL, and general HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis